CLINICAL TRIAL: NCT07124143
Title: The Effect of Platelet-Rich Plasma on Wound Healing After Gingivectomy: A Randomized Clinical Prospective Study
Brief Title: The Effect of Platelet-Rich Plasma on Wound Healing After Gingivectomy
Acronym: PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duygu Kilic (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Sponsor-Investigator, Duygu Kilic, Director, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 56733164/203
Record Dates: First submitted 2025-08-05; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Gingival Overgrowth
Keywords: gingival overgrowth; PRP; Gingivectomy; Wound Healing
MeSH Terms: conditions — Gingival Overgrowth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Control group) (No Intervention): Standard post-gingivectomy protocol without any agent applied to the surgical site
- Group 2 (Placebo) (Placebo Comparator): Standard protocol with 3-4 drops of physiological saline applied to the surgical site, four times a day, for 14 days.
  Interventions: Other: Placebo
- Group 3 (PRP Kit 1) (Active Comparator): Standard protocol with PRP prepared using Kit 1, applied to the surgical site in the same manner as the placebo group.
  Interventions: Other: PRP
- Group 4 (PRP Kit 2) (Active Comparator): Standard protocol with PRP prepared using Kit 2, applied to the surgical site in the same manner as the placebo group.
  Interventions: Other: PRP

INTERVENTIONS:
Other: PRP — venous blood will be drawn postoperatively and sent to Erciyes University Medical Faculty laboratories for PRP preparation. PRP will be centrifuged according to the manufacturer's specifications, transferred to sterile eye drop bottles, and given to the patients for application. Since PRP maintains its efficacy for seven days, a second blood draw and PRP preparation will be conducted during the first-week follow-up.
  Arms: Group 3 (PRP Kit 1); Group 4 (PRP Kit 2)
Other: Placebo — Patients will be provided with sterile eye drop bottles containing physiological saline and instructed to apply 3-4 drops to the wound site four times a day for 14 days.
  Arms: Group 2 (Placebo)

SUMMARY:
The aim of the study is to evaluate the effects of using droplet-form platelet-rich plasma (PRP), known to have positive effects during the intermediate healing process, on wound healing in areas left for secondary healing after gingivectomy.

After the gingivectomy procedure, patients will be divided into four groups, each consisting of 10 individuals:

Group 1 (Control Group): This group will follow the standard post-gingivectomy protocol without any agent applied to the surgical site.

Group 2 (Placebo Group): In this group, the standard protocol will be followed, and physiological saline will be applied to the surgical site in 3-4 drops, four times a day, for 14 days.

Groups 3 and 4 (Study Groups): These groups will follow the standard protocol, with PRP prepared using different kits applied to the surgical site in 3-4 drops, four times a day, for 14 days.

All patients in the groups will be evaluated on the 3rd, 7th, 14th, and 30th days after the gingivectomy procedure. Postoperative pain will be assessed using the Visual Analog Scale (VAS), while wound healing will be evaluated using the Healing Index (Landry et al.) based on photographs of the region. Before taking standardized photographs, the surgical area will be stained with two-tone dye.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effectiveness of platelet-rich plasma (PRP) prepared with different kits in improving the healing rate and enhancing patient comfort during the recovery process in the secondary healing areas following gingivectomy.

Systemically healthy individuals, patients with inflammatory gingival overgrowth, patients without periodontal treatment in the operative area within the last year, non-smokers and patients with intact periodontal structures will be included to the study. Also pregnant or breastfeeding patients, Patients below 18 or above 55 ages, smoking patients, patients with systemic diseases and who received periodontal treatment in the operative area within the last year and who use of medications causing gingival overgrowth will be excluded from the study.

Methodology:

A total of 40 patients meeting the inclusion criteria and willing to participate in the study will be recruited from those attending the Periodontology Clinic at Erciyes University Faculty of Dentistry for gum disease treatment.

Initial Procedures:

All participants will undergo initial periodontal treatment, including scaling and root planing. Periodontal assessments (plaque index, gingival index, probing depth, and attachment loss) will be performed before the initial treatment and at the first month post-treatment.

Study Procedure:

One month after the completion of initial periodontal therapy, gingivectomy will be performed, and the operative sites will be left for secondary healing. Before the procedure, the Pressure Pain Threshold Measurement will be taken for all patients using an algometer.

Participants will be randomly assigned to one of four groups:

Group 1 (Control group): Standard post-gingivectomy protocol without any agent applied to the surgical site.

Group 2 (Placebo): Standard protocol with 3-4 drops of physiological saline applied to the surgical site, four times a day, for 14 days.

Group 3 (PRP Kit 1): Standard protocol with PRP prepared using Kit 1, applied to the surgical site in the same manner as the placebo group.

Group 4 (PRP Kit2): Standard protocol with PRP prepared using Kit 2, applied similarly.

Postoperative Care:

All patients will be prescribed ibuprofen 600 mg (three times daily for three days). Placebo group patients will receive physiological saline in sterile eye drop bottles to apply as instructed.

In the PRP groups, venous blood will be drawn postoperatively and sent to Erciyes University Medical Faculty laboratories for PRP preparation. PRP will be centrifuged according to the manufacturer's specifications, transferred to sterile eye drop bottles, and given to the patients for application. Since PRP maintains its efficacy for seven days, a second blood draw and PRP preparation will be conducted during the first-week follow-up.

Follow-up and Assessments:

Patients will be evaluated on days 3, 7, 14, and 30 postoperatively. Pain assessment: Visual Analog Scale (VAS) will be used. Wound healing assessment: The surgical area will be stained with two-tone dye, standardized photographs will be taken, and the Healing Index (Landry et al.) will be used to evaluate healing on a 1-5 scale (1: very poor, 5: excellent).

At the one-month follow-up after gingivectomy, plaque index, gingival index, probing depth, and attachment loss measurements will be repeated.

This study aims to provide insights into the impact of PRP application on postoperative recovery and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals
* Patients with inflammatory gingival overgrowth
* Patients who have not received periodontal treatment in the area to be treated within the last year
* Non-smokers
* Patients with intact periodontal structures

Exclusion Criteria:

* Pregnancy or lactation
* Age under 18 or over 55
* Smoking
* Presence of systemic diseases
* Patients who have received periodontal treatment in the area to be treated within the last year
* Use of medications causing gingival overgrowth

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
The amount of wound healing | On the 3rd, 7th, 14th, and 30th days following the gingivectomy procedure
  The wound area was stained with two-tone dye, and standardized photographs will be taken. Wound healing then was evaluated using the Healing Index (Landry et al.) based on the photographs. The Healing Index is designed on a 1-5 scale, where 1 indicates very poor healing, and 5 indicates excellent healing.

SECONDARY OUTCOMES:
Periodontal changes | Before the initial periodontal treatment and at the first month after gingivectomy
  Plaque Index (PI): To determine the level of plaque accumulation.
postoperative pain | On the 3rd, 7th, 14th, and 30th days following the gingivectomy procedure
  Postoperative pain experienced by the patients was assessed using the Visual Analog Scale (VAS). An independent doctor assessed the pain score by using minimum 0, maximum 10 scores with 10-cm unscaled visual analog scale (VAS).
Periodontal changes | Before the initial periodontal treatment and at the first month after gingivectomy
  Gingival Index (GI): To assess gingival inflammation.
Periodontal changes | Before the initial periodontal treatment and at the first month after gingivectomy
  Clinical Attachment Loss (CAL): To evaluate the extent of attachment loss.
Periodontal changes | Before the initial periodontal treatment and at the first month after gingivectomy
  Probing Depth (PD): To measure the depth of periodontal pockets.

OTHER OUTCOMES:
Pressure Pain Threshold - PPT | Before the gingivectomy procedure
  An examiner touched the tip of the dial tension gauge perpendicular to the surface of the attached gingival mucosa at the midline of the maxilla and mandible. After a trial, the process was repeated three times with a 3-minute interval between measurements. The average of the three values was taken for statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Kılıç, Principal Investigator — Erciyes University Faculty of Dentistry Department of Periodontology
Locations (1):
- Erciyes University Faculty of Dentistry Department of Periodontology, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes